CLINICAL TRIAL: NCT02478723
Title: An Observational Study Evaluating the Sonendo GentleWave™ System and the EndoTechnologies CPoint™ Obturation for Treatment of Molar Teeth Requiring Root Canal Therapy
Brief Title: A Study Evaluating the Sonendo GentleWave™ System
Acronym: To The Point
Status: Terminated | Type: Observational
Why Stopped: Study device no longer manufactured by Sonendo. Total enrollment for the study was 20 subjects, only 3 subjects were enrolled and treated.
Sponsor: Sonendo, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CS-08
Record Dates: First submitted 2015-06-17; First posted 2015-06-23 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-03

CONDITIONS: Root Canal
Keywords: requiring therapy; Teeth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Sonendo GentleWave™ System — The Sonendo GentleWave System is intended to prepare, clean, and irrigate 1st and 2nd molar teeth indicated for root canal therapy.
  Other Names: EndoTechnologies CPoint™ Obturation

SUMMARY:
A post market, observational study evaluating the treatment of 1st and 2nd molars indicated for root canal therapy and treated with the Sonendo GentleWave System and obturated with CPoint and BC Sealer in at least one canal.

ELIGIBILITY:
Inclusion Criteria:

* The patient is 18 years of age or older
* The subject tooth has been treated for root canal therapy with the Sonendo GentleWave System and obturated with CPoint and BC Sealer in at least one canal
* The subject tooth is a 1st or 2nd molar

Exclusion Criteria:

* Vertical fracture, horizontal fracture, or perforation extending below the Cemento-Enamel Junction (CEJ) of the subject tooth
* Subject tooth having previous or attempted pulpectomy or root canal therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age or older, who have a 1st or 2nd molar tooth that received root canal therapy with the Sonendo GentleWave System and obturation with CPoint and BC Sealer in at least one canal.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-04 (Actual); Primary Completion 2018-01-24 (Actual); Study Completion 2019-03-27 (Actual)

PRIMARY OUTCOMES:
Subject teeth that are healed or are healing at the twenty-four month follow-up visit. | 24 months
  Healed is defined by absence of a radiographic indication of apical periodontitis (Periapical Index Score < 3) and absence of clinical signs and symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Miller, Study Director — Sonendo, Inc.
Locations (1):
- Sonendo, Laguna Hills, California, United States